CLINICAL TRIAL: NCT05185687
Title: Race, Status, Vaccines, Tests, and Place: Public Attitudes and Support for Equitable COVID-19 Vaccine and Test Allocation
Brief Title: Public Support for COVID-19 Test Allocation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Alison Buttenheim, Associate Professor of Nursing and Health Policy, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 848725; #84525 (Registry Identifier: AsPredicted)
Record Dates: First submitted 2022-01-07; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Health Equity; COVID-19
Keywords: Allocation of Healthcare Resources
MeSH Terms: conditions — COVID-19 | interventions — Random Allocation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First Come, First Served (Experimental): Respondents will view the following description: "The US government will make 500 million COVID-19 home tests available for free. US residents can ask for tests by entering their home address in a website. It is likely that more people will want tests than will be available. How should the government decide who will receive tests, when there are not enough for all who want them? One plan that is being considered is this one:"
  Below this statement, respondents will view the "First Come, First Served" plan description.
  Interventions: Behavioral: First Come, First Served
- Random (Experimental): Respondents will view the following description: "The US government will make 500 million COVID-19 home tests available for free. US residents can ask for tests by entering their home address in a website. It is likely that more people will want tests than will be available. How should the government decide who will receive tests, when there are not enough for all who want them? One plan that is being considered is this one:"
  Below this statement, respondents will view the "Random" plan description.
  Interventions: Behavioral: Random
- Disadvantaged Priority & Random (Experimental): Respondents will view the following description: "The US government will make 500 million COVID-19 home tests available for free. US residents can ask for tests by entering their home address in a website. It is likely that more people will want tests than will be available. How should the government decide who will receive tests, when there are not enough for all who want them? One plan that is being considered is this one:"
  Below this statement, respondents will view the "Disadvantaged Priority & Random" plan description.
  Interventions: Behavioral: Disadvantaged Priority & Random

INTERVENTIONS:
Behavioral: First Come, First Served — Respondents will view the following description of the plan: "Tests will be sent out in the order they are requested. People who request tests the quickest will get them first, no matter where they live. People who request tests later may not get any. This strategy is also known as 'First Come, First Served.'"
  Arms: First Come, First Served
Behavioral: Random — Respondents will view the following description of the plan: "People who request tests will be entered into a random drawing, like a sweepstakes or lottery. Everyone who is in the drawing has the same chance of getting tests, no matter where they live, but some people may not get any tests."
  Arms: Random
Behavioral: Disadvantaged Priority & Random — Respondents will view the following description of the plan: "Because COVID-19 has hit people living in disadvantaged areas of the country harder, a proportion of tests will be sent exclusively to people in these zip codes. Planners will allocate 80% of the tests using a random drawing, like a sweepstakes or lottery. Everyone who is in the drawing has the same chance of getting tests, no matter where they live. The remaining 20% are set aside exclusively for the most disadvantaged areas, again allocated with a random drawing. Some people may not get any tests. But people living in disadvantaged areas are more likely to get them."
  Arms: Disadvantaged Priority & Random

SUMMARY:
In a randomized survey experiment, investigators will assess public support or opposition towards one of three potential government plans for allocating at-home coronavirus disease 2019 (COVID-19) tests to United States residents: 1) first come, first served; 2) a random draw; or 3) a random draw with 20% of tests reserved for disadvantaged areas. Investigators will also examine public attitudes surrounding other logistical and equity-related aspects of these allocation plans.

DETAILED DESCRIPTION:
Complementing other efforts to increase access to COVID-19 testing in the United States, the federal government recently announced the purchase of 500,000,000 at home COVID-19 to be distributed for free "to Americans that want them". A central logistical element in matching supply with demand will be a website, on which people will register their interest in getting tests delivered to their home address. However, it is still unclear how supply will be matched with demand. Three main candidate options are first come, first served (FCFS), in which people are sent tests in the order in which they make requests; a random draw, such as a lottery; or a combination of a random draw with a guaranteed reserved amount for more disadvantaged populations. FCFS is a widely known and practiced rationing principle, but it has shown to exacerbate inequities in, for example, the allocation of vaccine appointments. Random draws can mitigate this impact, but, in the present context, might be insufficiently sensitive to the fact that not everyone has internet access, and that the need for testing is greater among more disadvantaged communities. Combining a lottery with a disadvantage reserve system using measures such as the CDC's Social Vulnerability Index is a practical way of promoting equity, and it was already used by the majority of US states in allocating vaccines. The main objective of this study is to assess public support for each of these three allocation plans and describe differences by demographic characteristics. Investigators will also assess public attitudes toward specific details of these allocation plans. The study, which is expected to take approximately 5 minutes to complete, will be administered as part of an omnibus online survey.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or older, United States resident

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2019 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Support for allocation plan | 5 minutes
  Self-reported degree of support for the plan, measured on a 5-point Likert scale ("strongly oppose" to "strongly support") that will be collapsed into 3 response categories ("oppose," "neutral," and "support") for analysis.

SECONDARY OUTCOMES:
Household-level test allocation preference | 5 minutes
  Preferred way of sending tests to households, measured as a binary choice between a fixed or variable (based on household size) number of tests per household.
Tests allocated to disadvantaged areas | 5 minutes
  Self-reported percentage of tests wanted to be sent to disadvantaged areas, measured as a continuous variable on a slider from 0% to 100% with increments of 0.1%. This outcome will only be measured for respondents in the "Disadvantaged Priority & Random" condition.

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Buttenheim, PhD, MBA, Principal Investigator — University of Pennsylvania
Locations (1):
- Harris Insights & Analytics, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only de-identified individual participant data will be shared by Harris Insights & Analytics to the research team. Each participant will have a unique identifier to protect their confidentiality. Only authorized research personnel will have access to the data which will be maintained on encrypted hard-drives. Individual participant data may be made available to other researchers in an open-access repository.